CLINICAL TRIAL: NCT00671567
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Outpatient, Safety and Efficacy Study of TAK-375 in Adults With Chronic Insomnia
Brief Title: Ramelteon in Adults With Chronic Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-02-TL-375-020; U1111-1114-3130 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Insomnia
Keywords: Sleep Disorder; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 16 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon, 8 mg, tablets, orally, once daily for up to 5 weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Ramelteon — Ramelteon, 16 mg, tablets, orally, once daily for up to 5 weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 16 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once daily for up to 5 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Ramelteon, once daily (QD), in adult subjects with chronic insomnia.

DETAILED DESCRIPTION:
Insomnia is characterized by difficulties initiating and maintaining sleep or complaints of nonrestorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had "ever had difficulty sleeping." Based on reports of "regular" or "frequent" sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is a melatonin-1 receptor agonist under global development by Takeda Chemical Industries, Ltd, for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

This study is designed to determine the safety and efficacy of 35-day treatment of chronic insomnia with Ramelteon, using subjective measures of sleep. Total subject participation time in this study is expected to be approximately 2 months.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Has had primary insomnia as defined by the Diagnostic and Statistical Manual of Mental Disorders, Text Revision and a history of daytime complaint(s) associated with disturbed sleep.
* Subjective sleep latency greater than or equal to 45 minutes and a subjective total sleep time less than or equal to 6.5 hours per night for at least 3 nights during the week of the lead-in period, based on subject diary.
* Habitual bedtime is between 8:30 PM and 12:00 AM.
* Body mass index between 18 and 34, inclusive.

Exclusion Criteria

* Known hypersensitivity to Ramelteon or related compounds, including melatonin.
* Previously participated in a study involving Ramelteon.
* Participated in any other investigational study, and/or taken any investigational drug within 30 days or five half-lives prior to the first day of single-blind study medication, whichever is longer.
* Sleep schedule changes required by employment (eg, shift worker) within three months prior to the first day of single-blind study medication, or has flown across greater than three time zones within seven days prior to screening.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to the first day of single-blind study medication.
* Has ever had a history of seizures, sleep apnea, chronic obstructive pulmonary disease, restless leg syndrome, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* History of psychiatric disorder (including anxiety or depression) within the past 12 months.
* History of drug addiction or drug abuse within the past 12 months.
* History of alcohol abuse within the past 12 months.
* Current significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic or metabolic disease unless currently controlled and stable with protocol-allowed medication 30 days prior to the first day of single-blind study medication.
* Uses tobacco products during nightly awakenings.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel.
* Any additional condition that in the Investigator's opinion would:

  * Affect sleep-wake function
  * Prohibit the subject from completing the study
  * Not be in the best interest of the subject.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * melatonin or other drugs or supplements known to affect sleep/wake function.
  * anxiolytics
  * hypnotics
  * antidepressants
  * anticonvulsants
  * sedating H1 antihistamines
  * systemic steroids
  * respiratory stimulants and decongestants
  * over-the-counter and prescription stimulants
  * over-the-counter and prescription diet aids
  * central nervous system active drugs (including herbal preparations with central nervous system effects)
  * narcotic analgesics
  * beta blockers
  * melatonin
  * St. John's Wort
  * kava-kava
  * gingko biloba

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 848 (Actual)
Dates: Start 2002-12; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Mean Subjective Sleep Latency per subject diary, from Nights 1 through 7 of double-blind treatment. | Weeks 1, 2, 3, 4, and 5 or Final Visit

SECONDARY OUTCOMES:
Mean Subjective Sleep Latency per subject diary, over the week preceding the Day 15, Day 22, Day 29, and Day 36 Visits. | Weeks 2, 3, 4, and 5 or Final Visit
Subjective Total Sleep Time | Weeks 1, 2, 3, 4, and 5 or Final Visit
Subjective Number of Awakenings. | Weeks 1, 2, 3, 4, and 5 or Final Visit
Subjective Ease of Falling Back to Sleep after Awakening. | Weeks 1, 2, 3, 4, and 5 or Final Visit
Subjective Sleep Quality. | Weeks 1, 2, 3, 4, and 5 or Final Visit
Clinician's Clinical Global Impression | Weeks 1, 2, 3, 4, and 5 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Science, Study Director — Takeda
Locations (70):
- United States (70):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tempe, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Chula Vista, California
  - Irvine, California
  - La Mesa, California
  - Newport Beach, California
  - Northridge, California
  - Oakland, California
  - Redlands, California
  - Spring Valley, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Clearwater, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Longwood, Florida
  - Pembroke Pines, Florida
  - Safety Harbor, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Blairsville, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Danville, Indiana
  - Evansville, Indiana
  - Shawnee Mission, Kansas
  - Bethesda, Maryland
  - Brockton, Massachusetts
  - Detroit, Michigan
  - Hattiesburg, Mississippi
  - St Louis, Missouri
  - Lawrenceville, New Jersey
  - Moorestown, New Jersey
  - Albuquerque, New Mexico
  - Mineola, New York
  - Williamsville, New York
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Altoona, Pennsylvania
  - Jenkintown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sellersville, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Johnson City, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Virginia Beach, Virginia
  - Gig Harbor, Washington

REFERENCES:
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI